CLINICAL TRIAL: NCT05556980
Title: Randomized Controlled Trial Comparing the Outcomes of Totally Laparoscopic Distal Gastrectomy and Laparoscopy-assisted Gastrectomy for Gastric Cancer
Brief Title: Totally Laparoscopic Distal Gastrectomy for Gastric Cancer
Acronym: TLDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Liu (Other)
Responsible Party: Sponsor-Investigator, Liu Liu, Clinical professor, The First Affiliated Hospital of University of Science and Technology of China
Organization: The First Affiliated Hospital of University of Science and Technology of China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLDG
Record Dates: First submitted 2022-09-18; First posted 2022-09-27 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Complications
Keywords: laparoscopy-assisted gastrectomy; totally laparoscopic gastrectomy; distal gastroectomy; postoperative hospital stay; survival; complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the Outcomes Assessor would not know which approach the patient received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- totally laparoscopic distal gastrectomy (Experimental): patients in this arm will receive totally laparoscopic distal gastrectomy
  Interventions: Procedure: totally laparoscopic distal gastrectomy
- laparoscopy-assisted distal gastrectomy (No Intervention): patients in this group will receive laparoscopy-assisted distal gastrectomy

INTERVENTIONS:
Procedure: totally laparoscopic distal gastrectomy — all the surgical procedure would be finished under laparoscopy
  Arms: totally laparoscopic distal gastrectomy

SUMMARY:
This study was designed as a randomized clinical trial comparing the totally laparoscopic distal gastrectomy with laparoscopy-assisted distal gastroectomy for patients with gastric cancer, in terms of short-term and long-term outcomes.

DETAILED DESCRIPTION:
When one patient was enrolled, he will be randomly divided into experimental group (totally laparoscopic distal gastrectomy) or control group (laparoscopy-assisted distal gastrectomy). When he receives surgery, intraoperative parameters would be recorded. when the patient discharges, the routine follow-up would be regularly performed for the survival.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-80 years old, no gender limitation;
* primary gastric cancer and planed for distal gastrectomy;

Exclusion Criteria:

* patients with total or proximal gastrectomy;
* patients with distant metastasis.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative stay | about one week to one month from the finish of surgery
  the time from the finish of surgery to discharge

SECONDARY OUTCOMES:
Survival | 3 year
  the survival rate at the third year from the finish of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xubing Zhang, Hefei, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No
there is a plan to make individual participant data (IPD) available to other researchers.